CLINICAL TRIAL: NCT07298187
Title: The Effect of Head Position on the Optik Nerve Sheath Diameter in Patients During Thyroid Surgery
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ziya Kayadurmuş, RESEARCH ASSİSTANT DOCTOR, Istanbul University - Cerrahpasa
Other Study IDs: 1274724
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Cancer; Thyroid and Parathyroid Surgery; Thyroid Adenoma
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
THE EFFECT OF HEAD POSİTİON ON THE OPTİC NERVE SHEATH DİAMETER İN PATİENTS DURİNG THYROİD SURGERY

DETAILED DESCRIPTION:
Aim: In thyroidectomy surgery, the patient's head is placed in hyperextension and the patient is placed in a semi-sitting position to facilitate access to the surgical site. This position of the head causes a decrease in venous return or partial obstruction of venous return due to stretching of the neck veins. The aim of our study is to demonstrate the effect of surgical position on intracranial pressure by measuring the optic nerve sheath diameter (OSSD) using ultrasonography in patients undergoing thyroid surgery and to determine its correlation with post-operative headaches.

Material And Method: Our study was conducted prospectively and randomly in patients undergoing elective total thyroidectomy. Patients aged 18-65 with an ASA score of 1-2 and an operation time of less than 4 hours were included in our study. Patients were positioned in the semi-Fowler position with a 30° extension of the head. Bilateral OSSD surgical positioning was applied, and after ensuring haemodynamic stability for 5 minutes and at the end of the operation, measurements were taken twice using ultrasound, and the average was recorded. The Visual Analogue Scale (VAS) was used to assess postoperative pain intensity. Headache was assessed and recorded at 15 minutes, 30 minutes, 1 hour, 24 hours, 3 days, and 7 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65, with an ASA score between 1 and 2 according to the American Society of Anesthesiologists (ASA) physical status classification system
* whose surgery duration was expected to be less than 4 hours were included in our study.

Exclusion Criteria:

* liver failure
* kidney failure
* intracranial masses
* history of hydrocephalus,
* migraine
* chronic hypoxemia or hypercarbic lung disease
* additional heart disease
* hemodynamic insufficiency
* neurological and psychiatric diseases,
* glaucoma
* patients in whom ocular USG could not provide adequate images
* patients with pathological problems involving the eyelid and its surrounding area
* patients with diseases such as periorbital cellulitis
* patients with preoperative headache complaints
* patients with known diseases that could cause increased intracranial pressure
* patients who refused to participate in the study were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ISTANBUL UNIVERSITY-CERRAHPASA
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
OPTİC NERVE SHEATH DİAMETER | INTRAOPERATİVE PERİOD(FROM İNDUCTİON TO THE END OF SURGERY)
  CHANGE İN OPTİC NERVE SHEATH DİAMETER MEASURED BY ULTRASOUND BEFORE AND AFTER POSİTİONİNG DURİNG THYROİDECTOMY

SECONDARY OUTCOMES:
POSTOPERATİVE HEADACHE SEVERİTY (VISUAL ANALOG SCALE) | WİTHİN SEVEN DAYS AFTER SURGERY
  THE SEVERİTY OF POSTOPERATİVE HEADACHE WİLL BE ASSESSED USİNG A VİSUAL ANALOG SCALE. THE LOWEST POSSIBLE SCORE ON THE VISUAL ANALOG SCALE WAS 0, AND THE HIGHEST POSSIBLE SCORE WAS 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, FATİH, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE INDIVIDUAL PARTİCİPANT DATA WİLL NOT BE SHARED BECAUSE OF İNSTİTUTİONAL AND ETHİCAL RESTRİCTİONS